CLINICAL TRIAL: NCT01243814
Title: A Double-blind, Randomized, Placebo-controlled Study of the Relative Efficacy of a Single Dose of Hyaluronan in the Treatment of Osteoarthritis of the Ankle
Brief Title: A Double-blind RCT of a Single Dose of Hyaluronan in the Treatment of Osteoarthritis of the Ankle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry DeGroot, M.D. (Other)
Responsible Party: Henry DeGroot, M.D., Henry DeGroot
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: N08-429
Record Dates: First submitted 2010-11-18; First posted 2010-11-19 (Estimated); Last update posted 2012-03-20 (Estimated); Status verified 2010-11

CONDITIONS: Osteoarthritis
Keywords: hyaluronate; hyaluronic acid; viscosupplementation
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- supartz (Active Comparator): active intervention arm
  Interventions: Device: hyaluronate intra-articular injection
- saline injection (Placebo Comparator): placebo intervention arm
  Interventions: Device: placebo injection

INTERVENTIONS:
Device: hyaluronate intra-articular injection — joint injection in ankle with hyaluronate
  Other Names: Supartz
  Arms: supartz
Device: placebo injection — joint injection with saline solution for placebo
  Other Names: saline injection
  Arms: saline injection

SUMMARY:
To compare the therapeutic effect of single intra-articular injection of hyaluronate with a single intra-articular injection of normal saline (placebo) for osteoarthritis of the ankle.

DETAILED DESCRIPTION:
This study is a randomized, prospective, double-blind (blinded observer) , saline solution-controlled, parallel experimental design. The study device is SUPARTZ (Seikagaku Corporation, Tokyo, Japan) a brand of sodium hyaluronate.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible, subjects had to be at least 18 years old, not pregnant, and have pain and osteoarthritis of the ankle of at least stage 2 on the Kellgren and Lawrence scale.
* Their AOFAS score had to be 90 points or less out of a possible 100 points.
* Eligible subjects had to be willing to discontinue all pain medications and NSAIDs other than the rescue pain medications provided in the study.

Exclusion Criteria:

* Persons with systemic inflammatory condition or infection of the ankle or nearby soft tissues,
* an injection of steroid or surgery on the involved joint within 6 months,
* local cellulitis, rash, skin condition
* diabetic or neuropathic Charcot arthropathy,
* significant vascular insufficiency,
* current treatment with anticoagulants,
* lower extremity pain syndromes, sciatica, sprains, plantar fasciitis,
* significant ankle instability or malalignment,
* any known allergy to any of the components of either injection, known or suspected allergy to birds or bird products,
* disabling degenerative joint disease of the ipsilateral hip, knee or foot were ineligible for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2009-10; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
AOFAS score, difference from mean at 6 weeks and 12 weeks | 6 weeks 12 weeks
  American Orthopaedic Foot and Ankle score

CONTACTS AND LOCATIONS:
Overall Officials: Henry DeGroot, MD, Principal Investigator — Newton-Wellesley Hospital
Locations (1):
- The office of Dr. Henry DeGroot, Newton, Massachusetts, United States